CLINICAL TRIAL: NCT04461925
Title: Treatment of Coronavirus COVID-19 Pneumonia (Pathogen SARS-CoV-2) With Cryopreserved Allogeneic Multipotent Mesenchymal Stem Cells of the Placenta and Umbilical Cord
Brief Title: Treatment of Coronavirus COVID-19 Pneumonia (Pathogen SARS-CoV-2) With Cryopreserved Allogeneic P_MMSCs and UC-MMSCs
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Cell Therapy (Industry)
Collaborators: Kyiv City Clinical Hospital # 4 (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #4/24.04.2020
Record Dates: First submitted 2020-07-01; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: COVID-19 Pneumonia
Keywords: Placenta-derived MMSCs; i/v infusions
MeSH Terms: interventions — Anti-Bacterial Agents; Ceftriaxone; Azithromycin; Hormones; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Experimental: stem cells therapy + treatment in according with approved by Ukrainian Health Ministry COVID-19 clinical protocol Experimental Group 1: Subjects with severe COVID-19 pneumonia shall be received three infusions of cryopreserved allogeneic P-MMSCs (1 million cells/kg body weight) at 2-days intervals: Day "1", Day "4", Day "7".
  Control Group: treatment in according with approved by Ukrainian MoH COVID-19 clinical protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): On the basis conventional symptomatic treatment and supportive therapy, P-MMSCs were given at 1 million cells/kg body weight/ time, once every 3 days for a total of 3 times: Day "1", Day "4", Day "7".
  Interventions: Procedure: Placenta-Derived MMSCs; Cryopreserved Placenta-Derived Multipotent Mesenchymal Stromal Cells; Drug: Antibiotics; Drug: Hormones; Drug: Anticoagulant Therapy; Device: Оxygen therapy
- Control Group (Active Comparator): Conventional symptomatic treatments such as antibacterial (ceftriaxone, azithromycin), anticoagulants, hormones, oxygen therapy, mechanical ventilation and other supportive therapies
  Interventions: Drug: Antibiotics; Drug: Hormones; Drug: Anticoagulant Therapy; Device: Оxygen therapy

INTERVENTIONS:
Procedure: Placenta-Derived MMSCs; Cryopreserved Placenta-Derived Multipotent Mesenchymal Stromal Cells — i/v infusions
  Other Names: P-MMSCs
  Arms: Experimental group
Drug: Antibiotics — per os
  Other Names: ceftriaxone and azithromycin capsules
Drug: Hormones — a moderate amount of dexamethasone i/v
  Other Names: dexamethasone
Drug: Anticoagulant Therapy — Sub-Q
  Other Names: Еnoxaparin
Device: Оxygen therapy — Оxygen therapy, mechanical ventilation and other supportive therapies
  Other Names: Оxygen insufflation

SUMMARY:
Assessment of the clinical effects of infusions of cryopreserved allogeneic multipotent mesenchymal stem cells of the placenta and umbilical cord for COVID-19 patients with acute respiratory distress syndrome.

DETAILED DESCRIPTION:
Currently, cell-based therapy and especially stem cell therapy has become a promising therapeutic field, in which many see opportunities to cure incurable diseases. Severe respiratory consequences of the COVID-19, the disease caused by the novel SARS-CoV-2 coronavirus, have prompted urgent need for novel therapies.

Cell-based approaches, primarily using mesenchymal stem cells (MSCs), have demonstrated safety and efficacy in patients with the acute respiratory distress syndrome (ARDS) - common manifestation of cytokine storms, and the cause of death in many COVID-19 patients.

Mesenchymal stem cells are a powerful immunomodulator, they secrete many anti-inflammatory biologically active substances (cytokines) that reduce the inflammatory process in the lungs. Also mesenchymal stem cells secrete numerous growth factors that contribute to the recovery of not only the affected lung tissue but also other organs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged at 18 years (including) - 75 years old.
* Laboratory confirmation of SARS-CoV-2 infection by reverse-transcription polymerase chain reaction (RT-PCR) from any diagnostic sampling source.
* Pneumonia that is judged by X-ray imaging.

In accordance with any one of the following:

* dyspnea (RR ≥ 30 times / min);
* finger oxygen saturation ≤ 93% in resting state;
* arterial oxygen partial pressure (PaO2) / oxygen absorption concentration (FiO2) ≤ 300MMHG (if possible);
* invasive ventilation< 48 h.

Exclusion Criteria:

* Male or female, aged at <18 years and > 75 years old.
* Pregnancy, lactation and those who are not pregnant but do not take effective contraceptives measures.
* Patients with malignant tumor, other serious systemic diseases and psychosis.
* Patients who are participating in other clinical trials.
* Inability to provide informed consent or to comply with test requirements.
* Co-Infection of HIV, syphilis.
* Invasive ventilation > 48 h.
* Combined with other organ failure (need organ support).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-05-02 (Actual); Primary Completion 2021-05-02 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Changes of oxygenation index PaO2/FiO2, most conveniently the P/F ratio. | up to 28 days
  Improvement of pulmonary function. Arterial oxygen tension PaO2 (in mmHg)/fractional inspired oxygen FiO2 (expressed as a fraction, not a percentage), most conveniently the P/F ratio. The normal P/F ratio is ~ 400-500 mmHg (~55-65 kPa). P/F ratio <300mmHg - sign of Acute Respiratory Distress Syndrome (ARDS)
Changes in length of hospital stay | up to 28 days
  Length of Hospital Stay
Changes in mortality rate | up to 28 days
  Marker for efficacy of treatment

SECONDARY OUTCOMES:
Changes of С-reactive protein (CRP, mg/L) | At baseline, Day 1, Week 1, Week 2, Week 4, Week 8
  Infection biomarker. Serum CRP levels can be used for early diagnosis of pneumonia, patients with severe pneumonia had high CRP levels.
Evaluation of Pneumonia Improvement | At baseline, Day 1, Week 1, Week 2, Week 4, Week 8
  CT assessment of pulmonary lesions and lung tissue changes
Duration of respiratory symptoms (difficulty breathing, dry cough, fever, etc.) | At baseline, Day 1, Week 1, Week 2, Week 4, Week 8
  Indirect response to lung function
Peripheral blood count recovery time | At baseline, Day 1, Week 1, Week 2, Week 4, Week 8
  Degree of infection

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nemtinov, MD, Study Director — Institute of Cell Therapy
Locations (1):
- Institute of Cell Therapy, Kyiv, Ukraine